CLINICAL TRIAL: NCT04572178
Title: Cash Payment and Counseling for Quitting Smoking During Pregnancy
Brief Title: Cash Payment and Counseling During Pregnancy
Acronym: MARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Liselotte-Beutel-Foundation (Unknown); Ministry of Social Affairs, Integration and gender Equality (Unknown)
Responsible Party: Principal Investigator, Sabina Ulbricht, Prof. Dr., University Medicine Greifswald
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Unimed
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Pregnancy Related; Incentives
Keywords: Smoking cessation; Pregnancy; Incentives; Counseling; Cash payment
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cash payment and brief behavioral counseling (Experimental): The intervention consists of in person counseling and cash payment. The participants receive 25 Euro per week if they have succeeded in quitting smoking. Quitting smoking is evaluated by carbon monoxide measurements twice a week.
  Interventions: Behavioral: Cash payment and brief behavioral counseling

INTERVENTIONS:
Behavioral: Cash payment and brief behavioral counseling — The intervention consists of: (i) in person brief behavioral counseling, (ii) the evaluation of the smoking status using breath carbon monoxide, and (iii) cash payment of 25 Euro if the reading does not exceed a carbon monoxide value "3 ppm" ( ppm = parts per million) on two consecutive measurements per week. The intervention starts at the earliest in pregnancy week 15 and lasts until the delivery. If they relapse, the reward is not paid. However, in the following week they have the opportunity to quit smoking and being rewarded again.

SUMMARY:
Smoking during pregnancy has harmful effects on both mother and unborn child. Studies have shown that small rewards can help smokers to quit. In our current study, we ask how such rewards are most effective in supporting smoking cessation in pregnancy.

DETAILED DESCRIPTION:
We would like to include up to 15 pregnant women. Inclusion criteria are: (i) current pregnancy, between pregnancy week 15 and 23 and, (ii) current smoking of at least one cigarette per day. After an initial survey, the participating women are scheduled twice a week for counseling and evaluation of their smoking status.They will receive cash payment of 25 Euro if her carbon monoxide reading does not exceed the value "3", on two consecutive dates per week. A second survey will be conduced in pregnancy week 36 and a third survey, eight weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Current smoking, at least one cigarette per day
* Pregnancy, between pregnancy week 15 and 23

Exclusion Criteria:

* Inadequate language skills
* Cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 15 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Drop-out rate | Baseline up to pregnancy week 36
  Measure: Analyses of drop-out rate (%)

SECONDARY OUTCOMES:
Differences in number of cigarettes per day by self report | Baseline up to pregnancy week 36
  Measure: (n), paper pencil assessment (self-report)
Attempts to stop smoking by self report | Baseline up to pregnancy week 36
  Measure: (n), paper pencil assessment (self-report)
Attempts to stop smoking by carbon monoxide measurement | Baseline up to pregnancy week 36
  Measure: Carbon monoxide level <4 ppm (ppm= parts per million, device: piCObaby smokerlyzer)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Ulbricht, Prof. Dr., Principal Investigator — University Medicine Greifswald, Dep. Prevention Research and Social Medicine
Locations (1):
- Institute for Comunity Medicine, Department Prevention Research and Social Medicine, Greifswald, Germany

DOCUMENTS (1):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04572178/Prot_000.pdf